CLINICAL TRIAL: NCT01381718
Title: A Phase II Placebo-Controlled Trial of Modafinil to Improve Neurocognitive Deficits in Children Treated for a Primary Brain Tumor
Brief Title: Modafinil in Treating Children With Memory and Attention Problems Caused by Cancer Treatment for a Brain Tumor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: SCUSF 0901; SCUSF-0901 (Other: SunCoast CCOP Research Base); ACCL0922 (Other: Children's Oncology Network); 5U10CA081920-11 (NIH)
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Results first posted 2021-08-13 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2018-09

CONDITIONS: Brain and Central Nervous System Tumors; Cognitive/Functional Effects; Fatigue; Neurotoxicity; Psychosocial Effects of Cancer and Its Treatment
Keywords: childhood brain tumor; neurotoxicity; fatigue; cognitive/functional effects; psychosocial effects of cancer and its treatment
MeSH Terms: conditions — Central Nervous System Neoplasms; Fatigue; Neurotoxicity Syndromes | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Participants receive modafinil orally (PO) once daily (QD) on days 1-42.
  Interventions: Drug: modafinil
- Arm II (Placebo Comparator): Participants receive placebo PO QD on days 1-42.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: modafinil — Given PO
  Arms: Arm I
Other: placebo — Given PO
  Arms: Arm II

SUMMARY:
RATIONALE: Modafinil may help improve memory, attention, and fatigue caused by cancer treatment.

PURPOSE: This phase II randomized trial studies how well modafinil works in treating children with memory and attention problems caused by cancer treatment for a brain tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether a 6-week drug trial of modafinil, compared to placebo, is associated with improvement in neurocognitive function as defined by direct assessment of attention in children with cognitive impairment after treatment for a primary brain tumor.

Secondary

* Determine whether modafinil, compared to placebo, is associated with improved executive function, as assessed using the BRIEF executive function and hippocampal learning and executive function tasks from the CogState battery. Determine whether modafinil, compared to placebo, is associated with improved attention, as assessed by the Conners' (3rd Edition) 3 Parent Rating Scale (CPRS-3) - Short Form.
* Determine whether modafinil, compared to placebo, is associated with reduced fatigue as assessed using the PedsQL Multidimensional Fatigue Scale.
* Evaluate the safety of modafinil in this population.

OUTLINE: This is a multicenter study. Participants are randomized to 1 of 2 treatment arms.

* Arm I: Participants receive modafinil orally (PO) once daily (QD) on days 1-42.
* Arm II: Participants receive placebo PO QD on days 1-42. Participants complete a semi-automated, computerized cognitive-testing system (CogState) designed to assess psychomotor, attention/vigilance, memory, and other components of executive function by presenting different tasks, each with its own set of rules, at baseline and after completion of study therapy. Participants also complete the PedsQL Multidimensional Fatigue Scale (Peds QL-MFS).

Parents or legal guardians complete the PedsQL-MFS, the Conners Parent Reported Scale (CPR-3), and the Behavior Rating Inventory of Executive Function (BRIEF) at baseline and after completion of study therapy.

Clinical and/or research staff administer the Systematic Assessment for Treatment Emergency Events (SAFTEE), a semi-structured interview designed to elicit adverse events, at baseline and periodically during study.

After completion of study therapy, participants are followed up for 30 days.

ELIGIBILITY:
INCLUSION CRITERIA:

* Age ≥ 6 years and ≤ 18 years 10 months at the time of study entry (so that participants will be < 19 at the 6 week evaluation, which is the upper age limit for which the included instruments are valid).
* Diagnosis of a primary brain tumor treated with at least one of the following:

  1. neurosurgical resection of the brain tumor;
  2. cranial irradiation; or
  3. any chemotherapy to treat the brain tumor.
* Off-treatment and progression-free for at least 12 months and ≤ 14 years. Treatment cessation is defined as the final dose of chemotherapy, the last dose (fraction) of radiation or date of surgery, whichever occurred last.
* Parent/Legal Guardian and child able to read English or Spanish.
* Vision and hearing (eyeglasses and/or hearing aid permissible) sufficient for valid test administration and cooperation with examinations.
* Availability of a reliable parent or legal guardian who is willing and able to complete all of the outcome measures and fulfill the requirements of the study, including administration of medications and accompanying the participant to all study visits.
* Females of childbearing potential must have a negative pregnancy test result and must agree to use a medically acceptable method of contraception throughout the entire study period and for 30 days after the last dose of study drug.
* Childbearing potential is defined as girls who are >Tanner stage 2, except for those who have documented pan pituitary insufficiency or other hormonal state incompatible with pregnancy.
* Urine pregnancy tests are acceptable.

EXCLUSION CRITERIA:

* Off treatment > 14 years
* Inability to perform the testing procedure (for example, because of aphasia, motor deficits affecting the dominant hand, or IQ < 70)
* Known cardiac disorders including arrhythmias, hypertension requiring treatment or structural heart disease
* Diagnosis of narcolepsy, sick sinus syndrome, arrhythmia or prolonged QTc
* History of stroke or head injury associated with loss of consciousness within 12 months of registration
* History of grade 2 depression or anxiety or treatment with antidepressants, antipsychotics or MAO inhibitors within 30 days of registration
* Concurrent treatment with any medications or substances that are potent inhibitors or inducers of CYP3A4, hepatic enzyme inducing antiepileptic drugs (EIAEDs),or other drugs known to affect the metabolism of modafinil. Examples include but are not limited to itraconazole, ketoconazole, doxycycline, rifampin, St. John's wort, phenytoin, phenobarbital, diazepam, tricyclic antidepressants.
* If patients were previously taking, EIAEDs, they must be off for > 2 weeks prior to study enrollment.
* Treatment with other stimulant medications within 14 days of registration; however, a diagnosis of ADHD does NOT exclude a child from participation
* Participants with known hypersensitivity to modafinil, armodafinil or any of its components

Ages: 6 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 112 (Actual)
Dates: Start 2011-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey P. Krischer, MD, PhD, Study Chair — University of South Florida; Nicole J. Ullrich, MD, PhD, Study Chair — Boston Children's Hospital
Locations (60):
- United States (60):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Miller Children's Hospital, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Children's Hospital of Colorado; Saint Joseph Hospital, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - A. I. duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lee Memorial Health System, Fort Myers, Florida
  - University of Florida, Gainesville, Florida
  - Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic- Pensacola, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - SunCoast CCOP Research Base at the University of South Florida, Tampa, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - St. Luke's Mountain States Tumor Institute, Boise, Idaho
  - University of Illinois at Chicago, Chicago, Illinois
  - Riley Hospital for Children- Indiana University, Indianapolis, Indiana
  - Kosair Children's Hospital, Louisville, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Children's Hospital Boston, Boston, Massachusetts
  - CS Mott/University of Michigan, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi, Jackson, Mississippi
  - Children's Mercy Hospital and Clinics, Kansas City, Missouri
  - Saint Louis University / Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Saint Louis University Cancer Center, St Louis, Missouri
  - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - New York University Langone Medical Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Doernbecher Children's Hospital/ Oregoon Health Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I - Modafinil: Participants receive modafinil orally (PO) once daily (QD) on days 1-42.
  modafinil: Given PO
- Arm II - Placebo: Participants receive placebo PO QD on days 1-42.
  placebo: Given PO
Period: Overall Study
Arm/Group | Arm I - Modafinil | Arm II - Placebo
Started | 56 | 56
Completed | 51 | 43
Not Completed | 5 | 13
Not completed — Withdrawal by Subject | 2 | 5
Not completed — Lost to Follow-up | 3 | 5
Not completed — Toxicity, side effects or complications related to study | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Arm I - Modafanil: Participants receive modafinil orally (PO) once daily (QD) on days 1-42.
  modafinil: Given PO
- Total: Total of all reporting groups
Arm/Group | Arm I - Modafanil | Arm II - Placebo | Total
Number analyzed (Participants) | 56 | 56 | 112
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12.12 (2.92) | 12.7 (3.12) | 12.41 (3.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 31 | 58
  Male | 29 | 25 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 8 | 16
  Not Hispanic or Latino | 45 | 46 | 91
  Unknown or Not Reported | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 7 | 13
  White | 47 | 43 | 90
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5
BMI [Mean (Standard Deviation); unit: kg/m^2] | 22.66 (7.53) | 21.5 (6.55) | 22.08 (7.05)
Weight in kg [Mean (Standard Deviation); unit: Kg] | 49.68 (25.72) | 47.72 (20.96) | 48.7 (23.38)
Height in cm [Mean (Standard Deviation); unit: cm] | 143.93 (17.34) | 149.74 (39.03) | 146.84 (30.21)
Primary Cancer Diagnosis [Count of Participants; unit: Participants]
  Medulloblastoma PNET or ATRT | 22 | 29 | 51
  Pilocytic Astrocytoma (Grade 1) | 10 | 10 | 20
  Ependymoma | 7 | 3 | 10
  Germinoma or non-germinomatous germ | 4 | 3 | 7
  Astrocytoma (Grade 2) | 3 | 3 | 6
  Other | 4 | 4 | 8
  Craniopharygioma | 3 | 1 | 4
  Optic Pathway Tumor (optic nerve, chiasmatic optic tract) | 1 | 1 | 2
  Choroid plexus tumor (all grades) | 1 | 0 | 1
  Oligodendroglioma | 0 | 1 | 1
  Pinealoma (all grades) | 1 | 0 | 1
  Missing | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Age-Adjusted Scores at Week Six From Baseline in the Attention Task of the CogState Battery
Description: CogState Battery. CogState is a semi-automated, computerized cognitive testing system that was developed as a rapid and accurate test of cognitive function specifically for repeated assessment that is sensitive to the effects of medication in children over the age of 5 years and in adults from different language, cultural and socio-economic backgrounds. The CogState tasks to assess processing speed, visual attention, working memory and executive function were used. The CogState battery was administered in the following order: Detection Task, Identification Task, One Card Learning Task, One Back Task, and lastly, the Modified Groton Maze Learning Task. It was administered at baseline and 6 weeks. A positive change from baseline is an improvement. There is not a minimum or maximum since the value is reported as a z-score, but with the mean = 0 and the SD = 1, the range should be between -3 and 3.
Time Frame: Baseline and 6 weeks
Population: Decreased number of participants analyzed is because not all participants had a CogState score at 6 weeks
Measure: Mean (Standard Deviation); unit: Z Score
Arm/Group | Arm I - Modafinil | Arm II - Placebo
Number analyzed (Participants) | 50 | 42
Z Score | -0.16 (0.71) | 0.14 (1.06)

2. Secondary Outcome: Number of Reported Adverse Events (AEs)
Description: AEs gathered using SAFTEE (Systematic Assessment for Treatment Emergent Effects) and participant report on daily log.
Time Frame: 30 days post intervention
Measure: Number; unit: Adverse Events
Arm/Group | Arm I - Modafinil | Arm II - Placebo
Number analyzed (Participants) | 56 | 56
Adverse Events | 76 | 26

3. Secondary Outcome: Change in Working Memory Score at 6 Weeks From Baseline as Assessed on BRIEF
Description: Behavior Rating Inventory of Executive Function (BRIEF). The BRIEF is a behavior rating scale designed to assess executive functions in the home and school environments. The measure was selected to provide parent-reported outcomes of problems related to attention, memory and executive function that occur in everyday life. The instrument was utilized to measure the change in working memory, according to the parent's perspective only, from baseline to 6 weeks. Scores are linear transformations of raw scores into T scores (mean = 50, SD = 10); higher scores indicate greater difficulties. The baseline score was subtracted from the 6 week score. Positive change from baseline is an improvement. The total scale ranges from 0 to 172. A T score >60 on the BRIEF working memory subscale indicates cognitive impairment.
Time Frame: Baseline and 6 weeks
Population: Not all participants had a BRIEF score at 6 weeks
Measure: Mean (Standard Deviation); unit: T Score
Arm/Group | Arm I - Modafinil | Arm II - Placebo
Number analyzed (Participants) | 51 | 43
T Score | -4.1 (7.4) | -4.5 (9.2)

4. Secondary Outcome: Change in PedsQL Score at 6 Weeks From Baseline
Description: PedsQL is Pediatric Quality of Life Inventory Multi-dimensional Fatigue Scale. This scale is designed as a generic symptom-specific instrument to measure fatigue. Higher scores indicate fewer symptoms of fatigue. It was administered at baseline and 6 weeks. The score is the sum of the answers. The baseline score was subtracted from the 6 week score. A positive change indicates worsening. The scale total score range is from 0-72 for both the parent and patient reported instruments.
Time Frame: Baseline and 6 weeks
Population: Not all participants had a completed PedsQL at Week 6
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Arm I - Modafinil | Arm II - Placebo
Number analyzed (Participants) | 51 | 43
Scores on a scale
  Parent Rating | 11.3 (17.6) | 11.4 (15.9)
  Patient Rating | 9.3 (16.5) | 6.9 (16.6)

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: Complete and frequent monitoring for AEs was incorporated into the study using SAFTEE (Systematic Assessment for Treatment Emergent Effects developed by the National Institute of Mental Health. The final SAFTEE assessment will take place 30 days after the last dose of study agent.
  Participants will use the Study Medication Log, completed daily, to document any adverse events. Staff will review logs and compare to SAFTEE report.
Arm/Group | Arm I - Modafanil | Arm II - Placebo
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/56 | 1/56
Other Adverse Events (participants affected / at risk) | 34/56 | 12/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I - Modafanil (N=56) | Arm II - Placebo (N=56)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Fracture
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I - Modafanil (N=56) | Arm II - Placebo (N=56)
Headache (Nervous system disorders) | 12 (18) | 7 (9)
Insomnia (Psychiatric disorders) | 13 (16) | 3 (3)
Agitation (Psychiatric disorders) | 4 (4) | 2 (2)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No